CLINICAL TRIAL: NCT00885274
Title: A Randomized Controlled Trial Comparing Two Timing Regimens of Pico-salax for Colon Cleansing Prior to Colonoscopy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Assistant professor of Medicine, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Hookey Pico-Salax Timing
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Pico-Salax

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Split Dose (Experimental): Doses of Pico-Salax split: one dose administered the night prior to colonoscopy and the other dose administered the day of the procedure.
  Interventions: Drug: Split Dose Pico-Salax
- Traditional Dose (Active Comparator): Both doses of Pico-Salax taken the evening prior to colonoscopy.
  Interventions: Drug: Pico-Salax

INTERVENTIONS:
Drug: Pico-Salax — Both doses of Pico-Salax taken the evening prior to colonoscopy
  Arms: Traditional Dose
Drug: Split Dose Pico-Salax — One dose of Pico-Salax taken the evening prior to colonoscopy and the other the morning of the procedure.
  Arms: Split Dose

SUMMARY:
Pico-Salax is an osmotic and stimulant bowel cleansing agent used prior to colonoscopy. It is unknown whether splitting the doses (i.e. taking the second dose the morning of the colonoscopy) results in a better bowel cleansing, as research with other agents suggests this may be the case. This study aims to assess whether splitting the dose of Pico-Salax results in a better bowel cleansing than traditional dosing.

ELIGIBILITY:
Inclusion Criteria:

* colonoscopy indicated

Exclusion Criteria:

* congestive heart failure
* ascites
* renal failure
* hyponatremia
* previous intestinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
bowel cleansing assessed by the Ottawa Bowel Preparation Scale | day of colonoscopy

SECONDARY OUTCOMES:
patient tolerance of preparation | day of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Flemming JA, Vanner SJ, Hookey LC. Split-dose picosulfate, magnesium oxide, and citric acid solution markedly enhances colon cleansing before colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2012 Mar;75(3):537-44. doi: 10.1016/j.gie.2011.09.018. Epub 2011 Dec 21. PMID 22192423